CLINICAL TRIAL: NCT02869776
Title: Integrating HCV and HIV Screening During the Era of HIV Antigen Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-35271; RA25035163 -01A 1 (Other Grant/Funding Number: University of California, San Francisco); 5P30AI042853-18 (NIH)
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: HIV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Surveys and Questionnaires; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid finger stick (Experimental): HIV and HCV testing through rapid finger stick. Behavioral questionnaires will also be administered.
  Interventions: Behavioral: Questionnaire; Procedure: Rapid finger stick
- Standard venipuncture (Experimental): HIV and HCV testing through venipuncture. Behavioral questionnaires will also be administered.
  Interventions: Behavioral: Questionnaire; Procedure: Venipuncture

INTERVENTIONS:
Behavioral: Questionnaire — Behavioral questionnaires
Procedure: Rapid finger stick — HIV and HCV testing through rapid finger stick
  Arms: Rapid finger stick
Procedure: Venipuncture — HIV and HCV testing through venipuncture
  Arms: Standard venipuncture

SUMMARY:
The objective of this proposal is to develop an optimal testing strategy for HCV and HIV in high prevalence settings, such as detoxification centers with a large proportion of young injection drug users. The latest venipuncture testing will be compared to rapid finger stick testing for HCV and HIV. Outcomes for each strategy among individuals admitted at a short-term drug detoxification center will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18
* All clients admitted to BTC with a history of drug or alcohol use
* Individuals who self-report as being HIV and HCV non-infected within the past 6 months or having unknown status
* Participants providing contact information of two family members or friends
* Individuals signing a medical records release form for the referral site (Boston Medical Center)
* English speaking

Exclusion Criteria:

* Individuals unable to provide informed consent
* Individuals with a known history of HCV and/or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Number of participants who receive HCV test results | within 5 days (by the time of discharge from the detoxification center)
  The number of participants who receive HCV test results by the time they are discharged from the detoxification center
Number of participants who receive HIV test results | within 5 days (by the time of discharge from the detoxification center)
  The number of participants who receive HIV test results by the time they are discharged from the detoxification center

SECONDARY OUTCOMES:
Number of participants who link to HCV care | by three months
  The number of participants who are seen for an HCV visit
Number of participants who have HCV RNA testing | by three months
  The number of participants who have HCV RNA testing performed
Number of participants who have fibrosis staging performed | by three months
  The number participants who have fibrosis staging performed
Number of participants who have HCV treatment initiated | by six months
  The number participants who have HCV treatment initiated
Number of participants who reach sustained virologic response | by twelve months
  The number participants who reach sustained virologic response
Number of participants who link to HIV care | by 3 months
  The number participants who are seen for an HIV visit
Number of participants who HIV RNA testing | by 3 months
  The number participants who have HIV RNA testing
Number of participants who have CD4 testing | by 3 months
  The number participants who have CD4 testing
Number of participants who have antiretroviral treatment initiated | by 3 months
  The number participants who initiated antiretroviral treatment
Number of participants who achieve HIV viral suppression | by 6 months
  The number participants who achieve HIV viral suppression

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Assoumou, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Assoumou SA, Paniagua SM, Gonzalez P, Wang J, Beckwith CG, White LF, Taylor JL, Coogan K, Samet JH, Linas BP. HIV Pre-exposure Prophylaxis and Buprenorphine at a Drug Detoxification Center During the Opioid Epidemic: Opportunities and Challenges. AIDS Behav. 2021 Aug;25(8):2591-2598. doi: 10.1007/s10461-021-03220-0. Epub 2021 Mar 22. PMID 33751315
- [Derived] Assoumou SA, Paniagua SM, Linas BP, Wang J, Samet JH, Hall J, White LF, Beckwith CG. Rapid Versus Laboratory-Based Testing for HIV and Hepatitis C at a Drug Detoxification Treatment Center: A Randomized Trial. J Infect Dis. 2020 Sep 2;222(Suppl 5):S376-S383. doi: 10.1093/infdis/jiaa162. PMID 32877557